CLINICAL TRIAL: NCT01338376
Title: Organization Program of DiabEtes INsulIN ManaGement: An Open, Multi-center, Prospective, Randomized, 16-week, Controlled Clinical Study
Brief Title: Organization Program of DiabEtes INsulIN ManaGement
Acronym: OPENING
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Diabetes Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scilin20110124
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Education Group (Experimental): Subjects received structured diabetes education
  Interventions: Behavioral: Structured Education; Drug: Scilin®M30
- Conventional Care Group: (Active Comparator): Subjects received conventional diabetes education
  Interventions: Behavioral: Conventional Diabetes Education; Drug: Scilin®M30

INTERVENTIONS:
Behavioral: Structured Education — All of the educators who are responsible for the intensive group will be trained with the standard contents before the study kick-off.
  * Educator Activities: insulin injection, SMBG instruction, self-learned manuals, periodic assessment for subjects, subject counseling, self-care education (healthy eating, exercise, weight control), prevention and treatment of hypoglycemia complication education ,newsletter delivered by SMS
  * Physician Activity: frequent insulin titration
  Arms: Structured Education Group
Behavioral: Conventional Diabetes Education — The activities of the educators who are responsible for conventional group are identical with their routine clinical practice.
  * Educator Activities: insulin injection, SMBG instruction, healthy eating , prevention and treatment of hypoglycemia
  * Physician Activity: less frequent insulin titration
  Arms: Conventional Care Group:
Drug: Scilin®M30 — Subjects will be treated with Scilin®M30 twice daily

SUMMARY:
Diabetes is a common, costly condition associated with significant morbidity and mortality. Diabetes self-management education, the process of teaching individuals to manage their diabetes, has been considered an important part. The intensive education has the capacity to deliver effective interventions to a large number of people. The investigators may be able to redirect our efforts to diabetes care and education strategies that will have a positive impact on the optimization of glycemic control and the prevention of long-term complications of diabetes, reducing the subsequent human and health care costs.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, controlled clinical study. 1500 subjects with Type 2 DM will be enrolled and be randomized into Structured Education Group and Conventional Education Group in 1:1 ratio. Subjects in both of the groups will be treated with Scilin®M30 twice daily (30 minutes before breakfast and dinner). All the previous oral antidiabetic drugs (OAD(s)) will be discontinued except metformin and alpha-Glucosidase Inhibitors. The physician will determine the starting dose (0.3 IU/kg～0.4IU/kg), as well as later changes to dose according to insulin titration algorithm. The treatment duration will last 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent obtained before any trial-related activities Type 2 DM subjects;
* Age > 18 years old,male or female;
* Continuous treated with two or more oral antidiabetic drugs (OADs) for the last 3 months,and the current HbA1c>7.5%;
* Cooperative with structured management;

Exclusion Criteria:

* Subjects with type 1 diabetes;
* Gestational diabetes mellitus and other specific types DM;
* Those who are unwilling to sign in ICF;
* Subjects with repeated hypoglycemia;
* Subjects with BMI>30kg/m2;
* Impaired liver function,defined as alanine aminotransferase (ALAT)>= 2.5 or alkaline phosphatase (ALP)>= 2 times upper referenced limit times upper normal limit;
* Females of childbearing age who are pregnant, breast-feeding or have the intention of becoming pregnant or not using adequate contraceptive methods throughout the trial (adequate contraceptive measures as required by local law or practice);
* Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation;
* Any other clinically significant condition or major systemic diseases, including serious coronary heart disease, cardiovascular disease, myocardial infarction within the past 12 months; severe neurology or psychology or psychiatric diseases; serious infection; actively disseminated intravascular coagulation;
* Malignant neoplastic diseases (except carcinoma in situ);
* Current addiction to alcohol or other addictive substances;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Screen,16weeks
  Investigate glycemic control as measured by HbA1c change

SECONDARY OUTCOMES:
Assess diabetes self-management ability by Diabetes Management Self-Efficacy (C-DMSES) | Screen,16weeks
Diabetes self-management skills Diabetes self-management skills Assess diabetes self-care ability by Diabetes Self-Management (SDSCA) | Screen,16weeks
The satisfaction degree of structured management | Screen,2weeks,4weeks,8weeks,12weeks,16weeks
total daily insulin dose | 1week,2weeks,3weeks,4weeks,6weeks,8weeks,12weeks,16weeks
7-points of glucose | Screen,16weeks
  glucose before breakfast;glucose two hours after breakfast;glucose before lunch;glucose two hours after lunch;glucose before dinner;glucose two hours after dinner;glucose before sleep
body weight | baseline,2weeks,4weeks,8weeks,12weeks,16weeks
Medication compliance | Screen,16weeks
The incidence of Hypoglycemia | 1week,2weeks,3weeks,4weeks,6weeks,8weeks,12weeks,16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guo Xiao Hui, Professor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Guo XH, Ji LN, Lu JM, Liu J, Lou QQ, Liu J, Shen L, Zhang MX, Lv XF, Gu MJ. Efficacy of structured education in patients with type 2 diabetes mellitus receiving insulin treatment. J Diabetes. 2014 Jul;6(4):290-7. doi: 10.1111/1753-0407.12100. Epub 2013 Nov 26. PMID 24279284